CLINICAL TRIAL: NCT06090253
Title: A Hybrid Effectiveness-implementation Evaluation on Programs Promoting Healthy Aging With Sport Exercise (PHASE Program)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHASE
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ageing Well
Keywords: Ageing; Exercise; Community-dwelling; Functional Capacity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Active (Experimental): Gerotechnology enhanced multi-component exercise or Football training sessions.
  Interventions: Behavioral: Gerotechnology enhanced multi-component exercise; Behavioral: Football
- General community-dwelling aged cohort (Experimental): Gerotechnology enhanced multi-component exercise.
  Interventions: Behavioral: Gerotechnology enhanced multi-component exercise
- Geriatric symptoms (Experimental): Walking exercise and slow sports and exercise.
  Interventions: Behavioral: Walking exercise; Behavioral: Slow sports and exercise
- Chronic disease burden (Experimental): Walking exercise and slow sports and exercise.
  Interventions: Behavioral: Walking exercise; Behavioral: Slow sports and exercise
- Frail (Experimental): Elderly home gym training service.
  Interventions: Behavioral: Home-based exercise
- Control (No Intervention): No training session will be provided.

INTERVENTIONS:
Behavioral: Gerotechnology enhanced multi-component exercise — Intervention courses will be divided into 3 categories: Musculoskeletal training course, Neuromuscular and fall prevention training course, and cardiometabolic training course. The courses will be enabled by wearable technology, digital platform and visual display. Each of the courses will be 8 weeks in length (1 session per week), and 60 minutes per session.
  Arms: Active; General community-dwelling aged cohort
Behavioral: Home-based exercise — The proposed elderly home gym training services will be conducted by professional fitness instructors and tailor-made for the participants. 4 personal training sessions will be assigned (once per week, 45 to 60 minutes per session).
  Arms: Frail
Behavioral: Walking exercise — Two interventions will be provided: A) Walk-focused intervention, B) Disease-related walk intervention for participants with chronic diseases.
  Arms: Chronic disease burden; Geriatric symptoms
Behavioral: Slow sports and exercise — Participants will receive 10 training sessions (once or twice per week, 2 hours per session) conducted by professional fitness instructors. The training programs can be selected according to the participants' preference, including water exercises, stretching/fitness/gymnastics, slow walking/jogging, sports massage, Tai Chi, Yoga, etc.
  Arms: Chronic disease burden; Geriatric symptoms
Behavioral: Football — The Football Training Programme will be arranged (10 training sessions+1 game day per stage, 4 stages per season). held on artificial turf football pitch or indoor sport facilities in 5 regions
  Arms: Active

SUMMARY:
The goal of this clinical trial is to provide scientific evaluation on the effects of Promoting Healthy Aging with Sport Exercise (PHASE) Programs on the functional capacity of older. Based on the participants' mental well-being and physical health status, they will be provided with several tailored exercise intervention, including 1) football training; 2) gero-technology enhanced multi-component exercise; 3) slow sports and exercise; 4) walking exercise; 5) home-based exercise. A control group is also recruited and provided with no exercise intervention.

DETAILED DESCRIPTION:
This clinical trial is aimed to match a range of sport exercise to older adults who are in the different phase of transition along the continuum of intrinsic capacity, and to explore effective measures to promote healthy aging. The effectiveness of the tailored interventions will be tested among the six study arms of older adults with different intrinsic capacities, with five intervention arms and one control. Exercise intensity will be measured for each participant. The outcomes are overall health status, physical function, psychological function, and cognitive function. The outcomes are measured at baseline (pre-intervention), 3 months (post-intervention), and 6 months (post-intervention) to explore the program benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years

Exclusion Criteria:

* Any contraindication to exercise training

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1940 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Health status self-rated score | Changes from baseline to 3 month and 6 month post-intervention
  Measure by EQ05D-5L (range -0.59-1.0), higher score better quality of life
Mobility limitation score | Changes from baseline to 3 month and 6 month post-intervention.
  Measured by Short Physical Performance Battery (range 0-12), higher score better physical performance
Activity level | Changes from baseline to 3 month and 6 month post-intervention
  Measured by International Physical Activity Questionnaire.
Functional mobility score | Changes from baseline to 3 month and 6 month post-intervention
  Score measured by Life Space Assessment questionnaire (range: 0-120), higher score better performance
Sarcopenia risk score | Changes from baseline to 3 month and 6 month post-intervention
  Measured by Sarcopenia(SARC) questionnaire and calf circumference in unit of cm (range0-20), higher score higher risk of sarcopenia
Hand grip strength | Changes from baseline to 3 month and 6 month post-intervention
  Hand grip strength measured by hand-held dynamometer in unit of KG
Loneliness score | Changes from baseline to 3 month and 6 month post-intervention
  Measured by UCLA Loneliness Scale questionnaire (range20-80), higher score greater loneliness
Cognitive function score | Changes from baseline to 3 month and 6 month post-intervention
  Measured by Montreal Cognitive Assessment (range 0-30), A score of 26 or over is considered to be normal.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided